CLINICAL TRIAL: NCT02478671
Title: Magnetic Resonance Imaging (MRI) to Assess Radial Artery Compression and Arterial Perfusion While TR Band is Applied
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo Medical Corporation (Industry)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TIS2015-002
Record Dates: First submitted 2015-05-19; First posted 2015-06-23 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Poor Peripheral Perfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TR Band (Experimental): Each subject will have a Terumo TR Band applied to the wrist with MRI scans done at differing band pressure levels. The diameter of the radial artery will be measured at each level of band compression.
  Interventions: Device: TR Band

INTERVENTIONS:
Device: TR Band — The radial artery will be compressed using a Terumo TR Band and artery diameter and perfusion will be measured

SUMMARY:
Subjects' radial artery diameters and plethysmography waveforms will be recorded by MRI and pulse oxymetry at varying levels of radial artery compression by the Terumo TR Band.

DETAILED DESCRIPTION:
In this study, the diameter of each subjects' radial artery will be measured using MRI imagery at varying degrees of radial artery compression by adjusting the amount of air injected into a Terumo TR Band. In addition, using pulse oxymetry, the perfusion waveform will be measured and recorded also while the subjects have a TR Band in place on their wrists.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male adult (has reached the legal majority age).
2. Subject has provided his/her written informed consent to participate in the trial prior to any study -related procedure being conducted.

Exclusion Criteria:

1. Abnormal result of either baseline Barbeau or reverse Barbeau tests.
2. Pregnant or breast feeding female.
3. Subject with contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Guimaraes, MD, Principal Investigator — Medical University of South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TR Band: MRI based radial artery measurement
Period: Overall Study
Arm/Group | TR Band
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TR Band
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 25 [24 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: MRI Based Radial Artery Measurement
Description: Each subject's radial artery will be measured using MRI at varying levels of pressure within the TR Band.
Time Frame: Subjects will be followed up to one week post procedure
Measure: Mean (Full Range); unit: millimeters
Arm/Group | TR Band
Number analyzed (Participants) | 4
millimeters | 1.35 [0 to 2.7]

2. Secondary Outcome: Hand Perfusion as Measured by Pulse Oxymetry Waveform
Description: pulse oxymetry waveform will be used to measure arterial perfusion
Time Frame: Subjects will be followed up to one week post procedure
Measure: Mean (Full Range); unit: percent saturated
Groups:
- TR Band: Pulse Oxymetry
Arm/Group | TR Band
Number analyzed (Participants) | 4
percent saturated | 50 [0 to 100]

ADVERSE EVENTS:
Time Frame: from time of procedure until 1 week post procedure
Arm/Group | TR Band
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TR Band (N=4)
Dizziness (Nervous system disorders) | 1 (1) — Subject experienced approximately 10 seconds of dizziness when getting up from the MRI scanner table after the scans were completed. Dizziness resolved with no intervention.

LIMITATIONS AND CAVEATS:
Single center study with small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall be permitted to publish the results of the Study in a manner that fairly and accurately sets forth the conclusions reached. The party seeking publication shall submit to SPONSOR for review a draft of the proposed publication at least thirty (30) days prior to submission of the draft for publication.